CLINICAL TRIAL: NCT02495376
Title: REDEFINE AYAO: Reducing Emotional Distress, Enhancing Function and Improving Network Engagement in Adolescent and Young Adult Oncology
Brief Title: Reducing Emotional Distress, Enhancing Function and Improving Network Engagement in Adolescent and Young Adult Oncology
Acronym: REDEFINEAYAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Cancer Society, Inc. (Other); Robert H. Lurie Cancer Center (Other)
Responsible Party: Principal Investigator, David Victorson, Associate Professor of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00093614
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Cancer
Keywords: YACS; cancer; MBSR
MeSH Terms: conditions — Neoplasms | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Group A participates in the first available MBSR course.
  Interventions: Behavioral: MBSR
- Group B (Active Comparator): Group B waits 16 weeks before participating in the MBSR course.
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: MBSR — Based primarily on the instruction of mindfulness meditation and yoga, MBSR is a group-based, 8-week program that was developed at the University of Massachusetts Stress Reduction Clinic under the direction of Jon Kabat-Zinn. MBSR is comprised of a structured, developmentally sequenced curriculum that uses a group format to experientially instruct participants in the practice of mindfulness meditation and mindful Hatha yoga. Each session includes different forms of meditation practice, such as cultivating awareness of thoughts, feelings and bodily sensations, and learning to incorporate this awareness during stressful emotional and/or physical life situations.
  Other Names: mindfulness based stress reduction

SUMMARY:
We propose to examine the effects of mindfulness based stress reduction (MBSR) on outcomes of health related quality of life, disease symptoms, and biological correlates of stress in a sample of young adults with cancer. The proposed work will serve as an essential foundation for launching a program of clinical stress reduction research with this traditionally underserved population and has the potential to lead to the discovery of specific, modifiable psychosocial, behavioral, and biological mechanisms from which to address the problem of health disparities with this group.

DETAILED DESCRIPTION:
Primary Objective Examine the feasibility and acceptability of MBSR with YACs. We hypothesize that MBSR will be feasible and acceptable with this population, which will be assessed through examination of response rate and study attrition variables.

Secondary Objectives

1. Evaluate the effects of MBSR on outcomes of health related quality of life and disease symptoms among YACs.
2. Explore the impact of different forms of eHealth maintenance support following the MBSR intervention (instructor-delivered, peer-delivered, no message) to help uphold intervention effects over time.
3. Compare intervention and control groups on changes in biologic measures of stress (blood pressure, pulse, salivary cortisol, CRP and IL-6 biomarkers) over a 32-week period.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of any cancer between ages 18-39
* Must have signed and dated informed consent form, which includes agreeing to study procedures
* Must be currently between 18-39 years of age
* Must be able to read, write, speak and understand English
* Must be able to perform basic activities of daily living
* Must be cognitively intact and free of serious psychiatric illness
* Must have the ability to use a touchscreen keypad on a tablet device
* Must be willing to commit to either the MBSR course or waitlist control condition
* Must be willing to commit to eHealth intervention maintenance conditions
* Must be willing to complete all assessments

Exclusion Criteria:

* Bedridden, or physical debilitation such that study participation would not be feasible or would create undue hardship
* History of diagnosed severe mental illness or hospitalization for chronic psychiatric reasons, as identified by referring physicians
* Regular user of mindfulness-based stress reduction or a similar mind-body therapy (e.g., yoga, meditation), which is defined as ≥ 3 times a week for the past 2 weeks

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
feasibility assessed through examination of response rate and study attrition variables | week 33
  feasibility assessed through examination of response rate and study attrition variables

SECONDARY OUTCOMES:
effects on health related quality of life accessed through online questionnaires | baseline and study weeks 8, 16, 24, and 32
  effects on health related quality of life accessed through online questionnaires
the impact of eHealth maintenance support accessed through text message response | weekly, for the 8 consecutive weeks after the MBSR course
  the impact of eHealth maintenance support accessed through text message response
compare between-group changes in biologic measures of stress accessed through biomarkers | baseline and study weeks 16 and 32
  compare between-group changes in biologic measures of stress accessed through

CONTACTS AND LOCATIONS:
Overall Officials: David E Victorson, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bleyer A. The adolescent and young adult gap in cancer care and outcome. Curr Probl Pediatr Adolesc Health Care. 2005 May-Jun;35(5):182-217. doi: 10.1016/j.cppeds.2005.02.001. No abstract available. PMID 15841070
- [Background] Bleyer A. Young adult oncology: the patients and their survival challenges. CA Cancer J Clin. 2007 Jul-Aug;57(4):242-55. doi: 10.3322/canjclin.57.4.242. PMID 17626120
- [Background] White PH. Access to health care: health insurance considerations for young adults with special health care needs/disabilities. Pediatrics. 2002 Dec;110(6 Pt 2):1328-35. PMID 12456953
- [Background] Kirchhoff AC, Lyles CR, Fluchel M, Wright J, Leisenring W. Limitations in health care access and utilization among long-term survivors of adolescent and young adult cancer. Cancer. 2012 Dec 1;118(23):5964-72. doi: 10.1002/cncr.27537. Epub 2012 Sep 24. PMID 23007632
- [Background] Crom DB, Lensing SY, Rai SN, Snider MA, Cash DK, Hudson MM. Marriage, employment, and health insurance in adult survivors of childhood cancer. J Cancer Surviv. 2007 Sep;1(3):237-45. doi: 10.1007/s11764-007-0026-x. PMID 18648974
- [Background] Callahan ST, Cooper WO. Uninsurance and health care access among young adults in the United States. Pediatrics. 2005 Jul;116(1):88-95. doi: 10.1542/peds.2004-1449. PMID 15995037
- [Background] Martin S, Ulrich C, Munsell M, Taylor S, Lange G, Bleyer A. Delays in cancer diagnosis in underinsured young adults and older adolescents. Oncologist. 2007 Jul;12(7):816-24. doi: 10.1634/theoncologist.12-7-816. PMID 17673613
- [Background] Burke ME, Albritton K, Marina N. Challenges in the recruitment of adolescents and young adults to cancer clinical trials. Cancer. 2007 Dec 1;110(11):2385-93. doi: 10.1002/cncr.23060. PMID 17918260
- [Background] Ferrari A, Montello M, Budd T, Bleyer A. The challenges of clinical trials for adolescents and young adults with cancer. Pediatr Blood Cancer. 2008 May;50(5 Suppl):1101-4. doi: 10.1002/pbc.21459. PMID 18360838
- [Background] Bleyer A. Older adolescents with cancer in North America deficits in outcome and research. Pediatr Clin North Am. 2002 Oct;49(5):1027-42. doi: 10.1016/s0031-3955(02)00035-4. PMID 12430624
- [Background] Mattson MR, Demshar RK, Daly BJ. Quality of life of young adult survivors of hematologic malignancies. Cancer Nurs. 2013 Mar-Apr;36(2):E1-7. doi: 10.1097/NCC.0b013e31824242dd. PMID 22293158
- [Background] Victorson D, Cella D, Wagner LI, Kramer L, Smith ML. Measuring quality of life in cancer survivors. In: Feuerstein M, ed. Handbook of cancer survivorship. New York, NY: Springer; 2007:79-112.
- [Background] Kwak M, Zebrack BJ, Meeske KA, Embry L, Aguilar C, Block R, Hayes-Lattin B, Li Y, Butler M, Cole S. Prevalence and predictors of post-traumatic stress symptoms in adolescent and young adult cancer survivors: a 1-year follow-up study. Psychooncology. 2013 Aug;22(8):1798-806. doi: 10.1002/pon.3217. Epub 2012 Nov 8. PMID 23135830
- [Background] Phillips-Salimi CR, Andrykowski MA. Physical and mental health status of female adolescent/young adult survivors of breast and gynecological cancer: a national, population-based, case-control study. Support Care Cancer. 2013 Jun;21(6):1597-604. doi: 10.1007/s00520-012-1701-7. Epub 2013 Jan 10. PMID 23306935
- [Background] Mor V, Malin M, Allen S. Age differences in the psychosocial problems encountered by breast cancer patients. J Natl Cancer Inst Monogr. 1994;(16):191-7. No abstract available. PMID 7999464
- [Background] Mor V, Allen S, Malin M. The psychosocial impact of cancer on older versus younger patients and their families. Cancer. 1994 Oct 1;74(7 Suppl):2118-27. doi: 10.1002/1097-0142(19941001)74:7+3.0.co;2-n. PMID 8087779
- [Background] Coccia PF, Altman J, Bhatia S, Borinstein SC, Flynn J, George S, Goldsby R, Hayashi R, Huang MS, Johnson RH, Beaupin LK, Link MP, Oeffinger KC, Orr KM, Pappo AS, Reed D, Spraker HL, Thomas DA, von Mehren M, Wechsler DS, Whelan KF, Zebrack BJ, Sundar H, Shead DA. Adolescent and young adult oncology. Clinical practice guidelines in oncology. J Natl Compr Canc Netw. 2012 Sep;10(9):1112-50. doi: 10.6004/jnccn.2012.0117. PMID 22956810
- [Background] Hall AE, Boyes AW, Bowman J, Walsh RA, James EL, Girgis A. Young adult cancer survivors' psychosocial well-being: a cross-sectional study assessing quality of life, unmet needs, and health behaviors. Support Care Cancer. 2012 Jun;20(6):1333-41. doi: 10.1007/s00520-011-1221-x. Epub 2011 Jul 1. PMID 21720746
- [Background] NCCAM Definition of Mind Body Medicine. 2011.
- [Background] Barnes PM, Bloom B, Nahin RL. Complementary and alternative medicine use among adults and children: United States, 2007. Natl Health Stat Report. 2008 Dec 10;(12):1-23. PMID 19361005
- [Background] Wong SY. Effect of mindfulness-based stress reduction programme on pain and quality of life in chronic pain patients: a randomised controlled clinical trial. Hong Kong Med J. 2009 Oct;15 Suppl 6:13-4. No abstract available. PMID 19801710
- [Background] Chiesa A, Serretti A. Mindfulness-based stress reduction for stress management in healthy people: a review and meta-analysis. J Altern Complement Med. 2009 May;15(5):593-600. doi: 10.1089/acm.2008.0495. PMID 19432513
- [Background] Ledesma D, Kumano H. Mindfulness-based stress reduction and cancer: a meta-analysis. Psychooncology. 2009 Jun;18(6):571-9. doi: 10.1002/pon.1400. PMID 19023879
- [Background] Bohlmeijer E, Prenger R, Taal E, Cuijpers P. The effects of mindfulness-based stress reduction therapy on mental health of adults with a chronic medical disease: a meta-analysis. J Psychosom Res. 2010 Jun;68(6):539-44. doi: 10.1016/j.jpsychores.2009.10.005. Epub 2009 Dec 9. PMID 20488270
- [Background] Kabat-Zinn J. Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. New York: Dell Publishing; 1990.
- [Background] Bishop SR, Lau M, Shapiro S, et al. Mindfulness: A Proposed Ooperational Definition. Clinical Psychology: Science and Practice. 2004 2004;11(3):230-241.
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Vollestad J, Sivertsen B, Nielsen GH. Mindfulness-based stress reduction for patients with anxiety disorders: evaluation in a randomized controlled trial. Behav Res Ther. 2011 Apr;49(4):281-8. doi: 10.1016/j.brat.2011.01.007. Epub 2011 Jan 27. PMID 21320700
- [Background] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193
- [Background] Schmidt S, Grossman P, Schwarzer B, Jena S, Naumann J, Walach H. Treating fibromyalgia with mindfulness-based stress reduction: results from a 3-armed randomized controlled trial. Pain. 2011 Feb;152(2):361-369. doi: 10.1016/j.pain.2010.10.043. Epub 2010 Dec 13. PMID 21146930
- [Background] Esmer G, Blum J, Rulf J, Pier J. Mindfulness-based stress reduction for failed back surgery syndrome: a randomized controlled trial. J Am Osteopath Assoc. 2010 Nov;110(11):646-52. PMID 21135196
- [Background] Gross CR, Kreitzer MJ, Thomas W, Reilly-Spong M, Cramer-Bornemann M, Nyman JA, Frazier P, Ibrahim HN. Mindfulness-based stress reduction for solid organ transplant recipients: a randomized controlled trial. Altern Ther Health Med. 2010 Sep-Oct;16(5):30-8. PMID 20882729
- [Background] Gross CR, Kreitzer MJ, Reilly-Spong M, Wall M, Winbush NY, Patterson R, Mahowald M, Cramer-Bornemann M. Mindfulness-based stress reduction versus pharmacotherapy for chronic primary insomnia: a randomized controlled clinical trial. Explore (NY). 2011 Mar-Apr;7(2):76-87. doi: 10.1016/j.explore.2010.12.003. PMID 21397868
- [Background] Carlson LE, Ursuliak Z, Goodey E, Angen M, Speca M. The effects of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients: 6-month follow-up. Support Care Cancer. 2001 Mar;9(2):112-23. doi: 10.1007/s005200000206. PMID 11305069
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress, and immune parameters in breast and prostate cancer outpatients. Psychosom Med. 2003 Jul-Aug;65(4):571-81. doi: 10.1097/01.psy.0000074003.35911.41. PMID 12883107
- [Background] Carlson LE, Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. Int J Behav Med. 2005;12(4):278-85. doi: 10.1207/s15327558ijbm1204_9. PMID 16262547
- [Background] Matousek RH, Dobkin PL, Pruessner J. Cortisol as a marker for improvement in mindfulness-based stress reduction. Complement Ther Clin Pract. 2010 Feb;16(1):13-9. doi: 10.1016/j.ctcp.2009.06.004. Epub 2009 Jul 4. PMID 20129404
- [Background] Matousek RH, Pruessner JC, Dobkin PL. Changes in the cortisol awakening response (CAR) following participation in mindfulness-based stress reduction in women who completed treatment for breast cancer. Complement Ther Clin Pract. 2011 May;17(2):65-70. doi: 10.1016/j.ctcp.2010.10.005. Epub 2010 Nov 26. PMID 21457893
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress and levels of cortisol, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. Psychoneuroendocrinology. 2004 May;29(4):448-74. doi: 10.1016/s0306-4530(03)00054-4. PMID 14749092
- [Background] Simkin-Silverman LR, Wing RR, Boraz MA, Meilahn EN, Kuller LH. Maintenance of cardiovascular risk factor changes among middle-aged women in a lifestyle intervention trial. Womens Health. 1998 Fall;4(3):255-71. PMID 9787651
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331
- [Background] Kirsch NL, Shenton M, Rowan J. A generic, 'in-house', alphanumeric paging system for prospective activity impairments after traumatic brain injury. Brain Inj. 2004 Jul;18(7):725-34. doi: 10.1080/02699050310001646161. PMID 15204332
- [Background] Subrahmanyam K, Greenfield P. Online communication and adolescent relationships. Future Child. 2008 Spring;18(1):119-46. doi: 10.1353/foc.0.0006. PMID 21338008
- [Background] Van den Bulck J. Adolescent use of mobile phones for calling and for sending text messages after lights out: results from a prospective cohort study with a one-year follow-up. Sleep. 2007 Sep;30(9):1220-3. doi: 10.1093/sleep/30.9.1220. PMID 17910394
- [Background] Brown J. A review of the evidence on technology-based interventions for the treatment of tobacco dependence in college health. Worldviews Evid Based Nurs. 2013 Aug;10(3):150-62. doi: 10.1111/wvn.12000. Epub 2013 Feb 19. PMID 23421669
- [Background] Woolford SJ, Barr KL, Derry HA, Jepson CM, Clark SJ, Strecher VJ, Resnicow K. OMG do not say LOL: obese adolescents' perspectives on the content of text messages to enhance weight loss efforts. Obesity (Silver Spring). 2011 Dec;19(12):2382-7. doi: 10.1038/oby.2011.266. Epub 2011 Aug 25. PMID 21869762
- [Background] Rotheram-Borus MJ, Tomlinson M, Gwegwe M, Comulada WS, Kaufman N, Keim M. Diabetes buddies: peer support through a mobile phone buddy system. Diabetes Educ. 2012 May-Jun;38(3):357-65. doi: 10.1177/0145721712444617. Epub 2012 Apr 30. PMID 22546740
- [Background] Norman CD, Yip AL. eHealth promotion and social innovation with youth: using social and visual media to engage diverse communities. Stud Health Technol Inform. 2012;172:54-70. PMID 22910502
- [Background] McDade TW, Williams S, Snodgrass JJ. What a drop can do: dried blood spots as a minimally invasive method for integrating biomarkers into population-based research. Demography. 2007 Nov;44(4):899-925. doi: 10.1353/dem.2007.0038. PMID 18232218
- [Background] Levine A, Zagoory-Sharon O, Feldman R, Lewis JG, Weller A. Measuring cortisol in human psychobiological studies. Physiol Behav. 2007 Jan 30;90(1):43-53. doi: 10.1016/j.physbeh.2006.08.025. Epub 2006 Oct 19. PMID 17055006
- [Background] Fuligni AJ, Telzer EH, Bower J, Cole SW, Kiang L, Irwin MR. A preliminary study of daily interpersonal stress and C-reactive protein levels among adolescents from Latin American and European backgrounds. Psychosom Med. 2009 Apr;71(3):329-33. doi: 10.1097/PSY.0b013e3181921b1f. Epub 2009 Feb 5. PMID 19196810
- [Background] Bankier B, Barajas J, Martinez-Rumayor A, Januzzi JL. Association between C-reactive protein and generalized anxiety disorder in stable coronary heart disease patients. Eur Heart J. 2008 Sep;29(18):2212-7. doi: 10.1093/eurheartj/ehn326. Epub 2008 Jul 4. PMID 18603621
- [Background] Bankier B, Barajas J, Martinez-Rumayor A, Januzzi JL. Association between anxiety and C-reactive protein levels in stable coronary heart disease patients. Psychosomatics. 2009 Jul-Aug;50(4):347-53. doi: 10.1176/appi.psy.50.4.347. PMID 19687175
- [Background] Bankier B, Barajas J, Martinez-Rumayor A, Januzzi JL. Association between major depressive disorder and C-reactive protein levels in stable coronary heart disease patients. J Psychosom Res. 2009 Mar;66(3):189-94. doi: 10.1016/j.jpsychores.2008.09.010. Epub 2008 Oct 9. PMID 19232230
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] O'Donovan A, Hughes BM, Slavich GM, Lynch L, Cronin MT, O'Farrelly C, Malone KM. Clinical anxiety, cortisol and interleukin-6: evidence for specificity in emotion-biology relationships. Brain Behav Immun. 2010 Oct;24(7):1074-7. doi: 10.1016/j.bbi.2010.03.003. Epub 2010 Mar 18. PMID 20227485
- [Background] Corwin EJ, Johnston N, Pugh L. Symptoms of postpartum depression associated with elevated levels of interleukin-1 beta during the first month postpartum. Biol Res Nurs. 2008 Oct;10(2):128-33. doi: 10.1177/1099800408323220. PMID 18829596
- [Background] Slavich GM, O'Donovan A, Epel ES, Kemeny ME. Black sheep get the blues: a psychobiological model of social rejection and depression. Neurosci Biobehav Rev. 2010 Sep;35(1):39-45. doi: 10.1016/j.neubiorev.2010.01.003. Epub 2010 Jan 18. PMID 20083138
- [Background] McDade TW. Development and validation of assay protocols for use with dried blood spot samples. Am J Hum Biol. 2014 Jan-Feb;26(1):1-9. doi: 10.1002/ajhb.22463. Epub 2013 Oct 15. PMID 24130128
- [Background] Adam TC, Hasson RE, Ventura EE, Toledo-Corral C, Le KA, Mahurkar S, Lane CJ, Weigensberg MJ, Goran MI. Cortisol is negatively associated with insulin sensitivity in overweight Latino youth. J Clin Endocrinol Metab. 2010 Oct;95(10):4729-35. doi: 10.1210/jc.2010-0322. Epub 2010 Jul 21. PMID 20660036
- [Background] Adam EK, Doane LD, Zinbarg RE, Mineka S, Craske MG, Griffith JW. Prospective prediction of major depressive disorder from cortisol awakening responses in adolescence. Psychoneuroendocrinology. 2010 Jul;35(6):921-31. doi: 10.1016/j.psyneuen.2009.12.007. Epub 2010 Jan 15. PMID 20079576
- [Background] Adam EK, Kumari M. Assessing salivary cortisol in large-scale, epidemiological research. Psychoneuroendocrinology. 2009 Nov;34(10):1423-36. doi: 10.1016/j.psyneuen.2009.06.011. Epub 2009 Jul 31. PMID 19647372
- [Background] Chang C-H, Cella D. Equating health-related quality of life instruments in applied oncology settings. Physical Medicine and Rehabilitation: States of the Art Reviews. 1997 1997;11(2):397-406.
- [Background] Hambleton RK. Principles and selected applications of Item Response Theory. In: Linn R, ed. Educational Measurement: Third Edition. New York: American Council on Education; 1989:147-200.
- [Background] Hambleton RK. Emergence of item response modeling in instrument development and data analysis. Med Care. 2000 Sep;38(9 Suppl):II60-5. doi: 10.1097/00005650-200009002-00009. PMID 10982090
- [Background] Gershon RC. Computer adaptive testing. J Appl Meas. 2005;6(1):109-27. PMID 15701948
- [Background] Gershon RC. The effect of individual differences variables on the assessment of ability for computerized adaptive testing, Northwestern University; 1996.
- [Background] Jacobsen PB, Davis K, Cella D. Assessing quality of life in research and clinical practice. Oncology (Williston Park). 2002 Sep;16(9 Suppl 10):133-9. PMID 12380963
- [Background] Cella D, Chang CH. A discussion of item response theory and its applications in health status assessment. Med Care. 2000 Sep;38(9 Suppl):II66-72. doi: 10.1097/00005650-200009002-00010. No abstract available. PMID 10982091
- [Background] McHorney CA, Cohen AS. Equating health status measures with item response theory: illustrations with functional status items. Med Care. 2000 Sep;38(9 Suppl):II43-59. doi: 10.1097/00005650-200009002-00008. PMID 10982089
- [Background] Ware JE Jr, Bjorner JB, Kosinski M. Practical implications of item response theory and computerized adaptive testing: a brief summary of ongoing studies of widely used headache impact scales. Med Care. 2000 Sep;38(9 Suppl):II73-82. No abstract available. PMID 10982092
- [Background] Lai J-S, Cella D, Choi S, Teresi JA, Hays RD, Stone AA. Developing a fatigue item bank for the Patient-Reported Outcomes Measurement Information System (PROMIS FIB version 1). Presented at the Meeting of the Survey Methods in Multicultural, Multinational, and Multiregional Contexts (3MC), Berlin, Germany. 2008.
- [Background] Research OoBaSS. Progress and promise in research on social and cultural dimensions of health: A research agenda. Bethesda, MD: National Institutes of Health; 2001.
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Revicki DA, Chen WH, Harnam N, Cook KF, Amtmann D, Callahan LF, Jensen MP, Keefe FJ. Development and psychometric analysis of the PROMIS pain behavior item bank. Pain. 2009 Nov;146(1-2):158-69. doi: 10.1016/j.pain.2009.07.029. Epub 2009 Aug 15. PMID 19683873
- [Background] Gershon RC, Cella D, Fox NA, Havlik RJ, Hendrie HC, Wagster MV. Assessment of neurological and behavioural function: the NIH Toolbox. Lancet Neurol. 2010 Feb;9(2):138-9. doi: 10.1016/S1474-4422(09)70335-7. No abstract available. PMID 20129161
- [Background] Gotay CC, Pagano IS. Assessment of Survivor Concerns (ASC): a newly proposed brief questionnaire. Health Qual Life Outcomes. 2007 Mar 13;5:15. doi: 10.1186/1477-7525-5-15. PMID 17352831
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Clements AD, Parker CR. The relationship between salivary cortisol concentrations in frozen versus mailed samples. Psychoneuroendocrinology. 1998 Aug;23(6):613-6. doi: 10.1016/s0306-4530(98)00031-6. PMID 9802131
- [Background] Kirschbaum C, Wolf OT, May M, Wippich W, Hellhammer DH. Stress- and treatment-induced elevations of cortisol levels associated with impaired declarative memory in healthy adults. Life Sci. 1996;58(17):1475-83. doi: 10.1016/0024-3205(96)00118-x. PMID 8622574
- [Background] Stanton AL, Bower JE, Low CA. Posttraumatic growth after cancer. In: Calhoun LG, Tedeschi RG, editors. Handbook of Posttraumatic Growth: Research and Practice. Mahwah: Lawrence Erlbaum Associates, Inc; 2006:138-175.
- [Background] McDade TW, Burhop J, Dohnal J. High-sensitivity enzyme immunoassay for C-reactive protein in dried blood spots. Clin Chem. 2004 Mar;50(3):652-4. doi: 10.1373/clinchem.2003.029488. No abstract available. PMID 14981035
- [Background] Williams SR, McDade TW. The use of dried blood spot sampling in the national social life, health, and aging project. J Gerontol B Psychol Sci Soc Sci. 2009 Nov;64 Suppl 1(Suppl 1):i131-6. doi: 10.1093/geronb/gbn022. Epub 2009 Feb 25. PMID 19244547
- [Background] Wyatt G, Sikorskii A, Rahbar MH, Victorson D, Adams L. Intervention fidelity: aspects of complementary and alternative medicine research. Cancer Nurs. 2010 Sep-Oct;33(5):331-42. doi: 10.1097/NCC.0b013e3181d0b4b7. PMID 20467309
- [Background] Victorson D, Hankin V, Polster R, McCurdy M, McGuire M, Brendler C. Reducing Symptoms of Anxiety for Men with Prostate Cancer on Active Surveillance and their Spouses: Initial Findings from a Randomized Clinical Trial. The Journal of Urology. 2010 2010;138(4):e180-e181.
- [Background] Hankin V. Mindfulness Based Stress Reduction in Couples Battling Multiple Sclerosis. Midwestern Psychological Association. 2008 2008;18th Annual Meeting:12.
- [Result] Eyberg S, Edwards D, Boggs S, Foote R. Maintaining the Treatment Effects of Parent Training: The Role of Booster Sessions and Other Maintenance Strategies. Clinical Psychology: Science and Practice. 1998 1998;5:544-554.
- See also: American Cancer Society I. Cancer in Teens and Young Adults: Not Much Improvement? Accessed on February 24, 2013. — http://acspressroom.wordpress.com/2012/01/06/cancer-in-teens-and-young-adults-not-much-improvement/